CLINICAL TRIAL: NCT00421681
Title: Exercise Adherence Among Older Adults With Osteoarthritis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National Institute on Aging (NIA) (NIH)
Responsible Party: Susan L. Hughes, DSW, Professor and Co-Director, Center for Research on Health and Aging, Institute for Health Research and Policy, University of Illinois Chicago
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: AG0075; 5R01AG023424 (NIH)
Record Dates: First submitted 2007-01-10; First posted 2007-01-12 (Estimated); Last update posted 2009-12-14 (Estimated); Status verified 2008-01

CONDITIONS: Osteoarthritis
Keywords: Aging; exercise; health behavior
MeSH Terms: conditions — Osteoarthritis; Motor Activity; Health Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): Treatment Arm A will develop tailored/negotiated contracts with the exercise instructor to maintain post intervention exercise adherence at home or in the community. Half of the participants in this "negotiated maintenance" arm will be randomly assigned to receive telephone calls to reinforce adherence and half will be assigned to a no telephone calls group.
  Interventions: Behavioral: Fit and Strong! Exercise Program
- B (Experimental): Treatment Arm B will be mainstreamed into an ongoing facility-based exercise program for post intervention exercise adherence. Persons in this "mainstream follow up" arm will be randomly assigned such that half will receive regular telephone reinforcement follow up and half will not.
  Interventions: Behavioral: Fit and Strong! Exercise Program

INTERVENTIONS:
Behavioral: Fit and Strong! Exercise Program — Fit and Strong! is an 8-week (24 sessions) multi-component exercise and health education intervention, including flexibility, aerobic conditioning, strength training, and group discussion/problem solving for lifestyle change. Following participation in Fit and Strong!, all study participants are randomly assigned to one of 2 maintenance treatment follow-up groups.

SUMMARY:
The purpose of this study is to assess the comparative effects of two different ways of enhancing long-term adherence to and benefits associated with participation in the evidence-based, Fit and Strong multi-component exercise intervention for older persons with lower extremity osteoarthritis.

DETAILED DESCRIPTION:
Osteoarthritis (OA) is the most common condition affecting older people today. It is the leading cause of disability among older people and its impact is projected to increase substantially with the aging of the U.S population from 43 million currently to 60 million by 2020.

Promising 2- and 6-month outcomes have recently been reported from a randomized trial of a multi-component exercise intervention targeted at older adults with lower extremity OA. The Fit and Strong intervention, developed and tested as part of the Midwest Roybal Center for Health Maintenance, coupled strength training and aerobic walking with health education for sustained behavior change. Improvements have been found in confidence in ability to exercise, confidence in ability to continue exercising over time, lower extremity stiffness, lower extremity pain, and 6-minute distance walk. Importantly, the average adherence rate in the people who participated in the exercise intervention at six months was twice that reported by controls.

The specific aims of this study are to use a multi-site randomized controlled clinical trial to replicate the Fit and Strong intervention and to test the comparative effectiveness of a negotiated/tailored follow-up maintenance strategy vs. a mainstreaming, facility-based maintenance strategy, both of which will be tested with and without telephone reinforcement as an enhancement.

All enrolled participants will participate in the 8-week Fit and Strong exercise program designed specifically for older adults with lower-extremity OA. Prior to the conclusion of Fit and Strong participants will be randomly assigned to one of two follow-up maintenance groups. There is no more than minimal risk associated with this program.

ELIGIBILITY:
Inclusion Criteria:

* 60 years of age or older
* Presence of osteoarthritis in the lower extremities (including hip, knee, ankle, feet and lower back) with an American College of Rheumatology functional class rating of I, II, or III
* No other contraindication from a personal physician for participation in fitness walking or low-impact aerobics and strength training
* Lack of moderate to severe cognitive impairment shown as assessed by the Short Portable Mental Status Questionnaire

Exclusion Criteria:

* Under 60 years of age
* Lack of osteoarthritis in the lower extremities
* Contraindication from a personal physician for participation in activities described above
* Presence of moderate to severe cognitive impairment as assessed by the Short Portable Mental Status Questionnaire
* Steroid injections in either knee or hip within previous six months
* Knee or hip surgery within previous six months
* Plans for total knee or hip replacement within the next year
* Rheumatoid arthritis or other system inflammatory arthritis
* Diabetes that is not under good control
* Current participation in a structured aerobic exercise program
* Participation in original trial of the Fit and Strong Program

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2003-10; Primary Completion 2008-09 (Estimated); Study Completion 2008-09 (Estimated)

PRIMARY OUTCOMES:
Maintenance of exercise behavior measured by CHAMPS (Community Healthy Activities Model Program For Seniors) | Baseline, 2 months, 6 months, 12 months, 18 months

SECONDARY OUTCOMES:
Changes in lower extremity strength (timed sit-stand test) | Baseline, 2 months, 6 months, 12 months, 18 months
Aerobic capacity (6 minute distance walk) | Baseline, 2 months, 6 months, 12 months, 18 months
Pain, stiffness, physical function subscales measured by WOMAC (Western Ontario and McMaster osteoarthritis index) | Baseline, 2 months, 6 months, 12 months, 18 months
Functional ability measured by GeriAIMS (Geriatric Arthritis Impact Measurement Scale) | Baseline, 2 months, 6 months, 12 months, 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Susan Hughes, DSW, Principal Investigator — Center for Research on Health and Aging , University of Illinois, Chicago
Locations (1):
- Center for Research on Health and Aging, Chicago, Illinois, United States

REFERENCES:
- [Background] Hughes SL, Seymour RB, Campbell R, Pollak N, Huber G, Sharma L. Impact of the fit and strong intervention on older adults with osteoarthritis. Gerontologist. 2004 Apr;44(2):217-28. doi: 10.1093/geront/44.2.217. PMID 15075418
- [Background] Hughes SL, Seymour RB, Campbell RT, Huber G, Pollak N, Sharma L, Desai P. Long-term impact of Fit and Strong! on older adults with osteoarthritis. Gerontologist. 2006 Dec;46(6):801-14. doi: 10.1093/geront/46.6.801. PMID 17169935
- [Derived] Seymour RB, Hughes SL, Campbell RT, Huber GM, Desai P. Comparison of two methods of conducting the Fit and Strong! program. Arthritis Rheum. 2009 Jul 15;61(7):876-84. doi: 10.1002/art.24517. PMID 19565560